CLINICAL TRIAL: NCT06460727
Title: Effects of Task Oriented Exercice Training on Static Versus Dynamic Surface on Functional Mobility and Balance in Children With Cerebral Palsy
Brief Title: Task Oriented Training on Static Versus Dynamic Surface on Balance in CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0776
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Cerebral Palsy
Keywords: task oriented exercise training; functional mobility; cerebral palsy; Balance
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: It will be Randomized control trial in which non probabilty convenient sampling will be used. Two groups of 6-12 age will be formed in which participants will be randomly divided. Group A will only receive task oriented exercise training on dynamic surface and group B will receive task oriented task training on static surface.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- task oriented exercise training on dynamic surface (Experimental): This group will be provided with task specific exercise training on dynamic surface in cerebral palsy. Following exercises will be performed in this group: Make the child bounce on swiss ball, reaching the toy with both hand kept over the head on platform swing, high sitting on swiss ball throwing ball with both hands, reaching the toy with one hand shifting the wait towards reaching side. Exercise will be conducted 3 times per week for 8 weeks, pre and post session functional mobility will be measured by functional mobility scale and balance will be measured by Time up and Go test
  Interventions: Other: task oriented exercise training on dynamic surface
- task oriented training on static surface (Experimental): This group will be provided with task specific exercise training on static surface in cerebral palsy. The children in this group will receive following TOET: Sit to stand from various cjair heights , standing and reaching indifferent directions for an object, Stepping forwards, backwards, and sideways onto blocks of various heights, walking forward , backward and sideways, Walking up and down stairs. Exercise will be conducted 3 times per week for 8 weeks, pre and post session functional mobility will be measured by functional mobility scale and balance will be measured by Time up and Go test
  Interventions: Other: task oriented exercise training on static surface

INTERVENTIONS:
Other: task oriented exercise training on dynamic surface — Following exercises will be performed in this group: Make the child bounce on swiss ball, reaching the toy with both hand kept over the head on platform swing, high sitting on swiss ball throwing ball with both hands, reaching the toy with one hand shifting the wait towards reaching side.
  Arms: task oriented exercise training on dynamic surface
Other: task oriented exercise training on static surface — The children in this group will receive following TOET: Sit to stand from various cjair heights , standing and reaching indifferent directions for an object, Stepping forwards, backwards, and sideways onto blocks of various heights, walking forward , backward and sideways, Walking up and down stairs
  Arms: task oriented training on static surface

SUMMARY:
Cerebral palsy (CP) is a disorder characterized by abnormal tone, posture and movement which are due to a non-progressive interference, lesion, or abnormality of the developing/immature brain . It is clinically categorized into four groups according to the predominant motor syndrome: extra-pyramidal or dys-kinetic, spastic quadriplegia and spastic diplegia. The purpose of this current study is to determine the effect of a selected task-oriented training on balance and functional mobility in children with cerebral palsy. This will be a randomized clinical trial, data will be collected from Elite Physio and Special children center from Faisalabad. Study will be conducted on 22 patients.

Inclusion criteria of this study is children who can walk with or without walking aids from age between 6 to 12 years old. Cerebral palsy children who has any musculoskeletal deformity in any of two limb, visual auditory, perceptual and auditory deficits, seizures or epilepsy , having botulinum toxin injections will be excluded.

Group A will be provided with task oriented exercise training on dynamic surface.

Group B will be provided with task oriented exercise training on static surface.Pre and post session balance and functional mobility will be assessed by Time up and Go scale and Functional Mobility scale.

DETAILED DESCRIPTION:
Flow diagram for study data collection procedure (According to CONSORT guidelines) in case of an RCT.All the referred patient will be assessed for the eligibility criteria. Guardians of the patient will be asked to sign the consent .All the screened participents will be randomly allocated into two groups.( Group A TOET on dynamic surface) , (Group B TOET on static surface)

Group A: Dynamic surface group:

This group will be provided with task specific exercise training on dynamic surface in cerebral palsy. Following exercises will be performed in this group: Make the child bounce on swiss ball, reaching the toy with both hand kept over the head on platform swing, high sitting on swiss ball throwing ball with both hands, reaching the toy with one hand shifting the wait towards reaching side. Exercise will be conducted 3 times per week for 8 weeks, pre and post session functional mobility will be measured by functional mobility scale and balance will be measured by Time up and Go test.

Group B: Static surface group:

This group will be provided with task specific exercise training on static surface in cerebral palsy. The children in this group will receive following TOET: Sit to stand from various cjair heights , standing and reaching indifferent directions for an object, Stepping forwards, backwards, and sideways onto blocks of various heights, walking forward , backward and sideways, Walking up and down stairs. Exercise will be conducted 3 times per week for 8 weeks, pre and post session functional mobility will be measured by functional mobility scale and balance will be measured by Time up and Go test

ELIGIBILITY:
Inclusion Criteria:

* Children with cerebral palsy
* Age between 6 to 12 years
* Children with GMFCS level I and II

Exclusion Criteria:

* CP children who has any musculoskeletal deformity in any of two limb
* Visual auditory, perceptual and auditory deficits, seizures or epilepsy
* Having botulinum toxin injections

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Functional Mobility scale | 8 weeks
  A child's functional mobility level in everyday life is defined by the FMS over a distance of 5 m, 50 m, and 500 m, which correspond to the home, school, and community settings, respectively. For each distance, an ordinal rating from 1 to 6 is assigned depending on the amount of assistance required for the child's mobility
Time Up and Go Test: | 8 Weeks
  Children with CP who are ambulatory will be evaluated for balance, anticipatory postural control, and functional mobility using the Timed Up and Go (TUG) test. It can distinguish between children with various CP subtypes and those at levels I-III of the Gross Motor.
  Function Classification System (GMFCS) based on their performance. The TUG is a responsive and reliable test

CONTACTS AND LOCATIONS:
Overall Officials: Hira latif, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zai W, Xu N, Wu W, Wang Y, Wang R. Effect of task-oriented training on gross motor function, balance and activities of daily living in children with cerebral palsy: A systematic review and meta-analysis. Medicine (Baltimore). 2022 Nov 4;101(44):e31565. doi: 10.1097/MD.0000000000031565. PMID 36343029
- [Background] Chaudhari S, BV RS. A study to compare the effect of task oriented training versus functional progressive resistance exercise strength training on gross motor functions in spastic diplegics. Int J Physical Educ Sports Health. 2020;7(5):24-302020.